CLINICAL TRIAL: NCT04720937
Title: Knowledge, Perception, Attitude and Responsibility of Dentists Regarding Child Physical Abuse in Some Governorates of Upper Egypt
Brief Title: Knowledge, Perception, Attitude and Responsibility of Dentists Regarding to Physical Child Abuse in Some Governorates of Upper Egypt
Status: Completed | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Reham Samy Elsaid Ahmed Sadek, General dentist, Minia University
Other Study IDs: 352
Record Dates: First submitted 2021-01-17; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2019-12

CONDITIONS: Child Abuse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No

SUMMARY:
Child abuse and neglect (CAN), child maltreatment, and child victimization are interchangeable terms that refer to a major public health problem confronting children and families. . This study Investigated dentists' level of knowledge, perception, attitude & responsibility regarding child physical abuse in some of Upper Egypt governorates

ELIGIBILITY:
Inclusion Criteria:

* Dentists who working in Egyptian Ministry of health &/ or private dental clinics &/ or centres in three governorates of Upper Egypt (Minia, Assuit & Sohag).
* Dentists with all dental academic degrees (Bachelor, diploma, master, doctoral & other post graduate degree).

Exclusion Criteria:

* Dentists who are working in any other governorates except (minia, Assuit & Sohag).
* Under graduated dental students

Age Groups: Child, Adult, Older Adult
Study Population: Dentists
Sampling Method: Non-Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
knowledge | 1 year
  questionnaire used to assess dentists' knowledge level to high and low knowledge levels
perception | 1 year
  questionnaire used to assess dentists' perception level into high, moderate and low perception
attitude | 1 year
  questionnaire used to assess dentists' attitude level into positive and negative attitude

CONTACTS AND LOCATIONS:
Locations (1):
- Reham, Minya, Egypt